CLINICAL TRIAL: NCT03354910
Title: Comparing the Effectiveness of House Calls and Peer Mentorship to Reduce Racial Disparities in Live Donor Kidney Transplantation
Brief Title: House Calls and Peer Mentorship
Acronym: HC+PM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Medical University of South Carolina (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, James Rodrigue, Professor of Psychology in the Department of Psychiatry, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2017P000521; PCORI 1609-36589 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2017-10-23; First posted 2017-11-28 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Chronic Kidney Disease; End-Stage Renal Disease
Keywords: Live Donor Kidney Transplantation; LDKT; Disparity; African American; Education; Patient Support
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — House Calls

STUDY DESIGN:
Intervention Model Description: Treatment assignments will be based on a computer-generated randomization scheme, stratified by age (<60 vs. ≥60 yrs old) and household income (<250% vs. ≥250% of federal poverty guidelines), since older and low-income patients are known to have lower LDKT rates a priori. Patients will be randomized into one of three treatment arms in a 1:3:3 fashion such that 54 Usual Care, 160 HC and 160 HC+PM patients will be enrolled. The study investigators and research assistants conducting the study assessments of patients will remain blinded to the treatment assignments. KT candidates will be informed of group assignment immediately after completing the Baseline assessment.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (No Intervention): All enrolled patients will receive Usual Care for transplant candidates at our two centers, which includes individual meetings with transplant providers, attendance at a patient group education session in the transplant center (focused on the specifics of the transplant experience), and a transplant education binder.
- Usual Care (UC) + House Calls (HC) (Active Comparator): Patients and their invited guests will be scheduled for one House Call. A house call is meeting done at a patient's home with transplant health educators facilitating a discussion on topics related to living kidney donation. Patients and guests also receive an information packet containing several brochures providing information about the living donation process, common concerns and misperceptions, and donation resources and information about our transplant center (e.g., copy of our quarterly newsletter, contact information). Patients in the group will also receive Usual Care, the regular education on living donation, provided as part of their routine transplant care.
  Interventions: Behavioral: House Call
- UC + HC + Peer Mentorship (Experimental): Patients in this condition will receive the Usual Care and the House Calls intervention as described previously. In addition, participants will receive access to a Peer Mentor trained by the National Kidney Foundation following their House Call.
  Interventions: Behavioral: House Call; Behavioral: Peer Mentorship

INTERVENTIONS:
Behavioral: House Call — 60 to 90 minute home based educational intervention which will be administered by a health educator.
  Arms: UC + HC + Peer Mentorship; Usual Care (UC) + House Calls (HC)
Behavioral: Peer Mentorship — A National Kidney Foundation Peer Mentor will be assigned to the participant to provide contact and support to study participants.
  Arms: UC + HC + Peer Mentorship

SUMMARY:
Live donor kidney transplantation (LDKT) offers the most optimal survival and quality of life benefit for those with late-stage chronic kidney disease. However, minorities, especially blacks, are much less likely to receive LDKT than whites. Given the shortage of deceased donor organs, interventions expanding access to LDKT are needed, particularly for minority patients. House Calls (HC), an educational intervention developed by this study's PI has been shown to be an effective program for raising rates of live donation, especially for black patients. While the HC program has shown outstanding results, participant feedback suggested that follow-up may provide even more benefits. Previous research suggests that peer mentorship (PM) from former or current patients with ESRD may be effective in raising rates of living donation. As such, peer mentorship programs may act as an effective follow-up for HC participants. This study will examine the impact of the HC intervention combined with the peer mentorship program of the National Kidney Foundation on rates of live donor kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Black race (including possible Cape Verdean, Haitian, Dominican)
* ≥18 yrs old
* English speaking
* Meets eligibility criteria for kidney transplant evaluation
* Ability to provide informed consent
* Resides within 1.5 hr drive of HC educator

Exclusion Criteria:

* Temporarily Unavailable (TU) on the waiting list and TU is likely to exceed 6 months based on judgement of kidney transplant team
* Awaiting combined kidney-liver transplantation
* Awaiting simultaneous pancreas-kidney transplantation
* Participation in another study to increase the likelihood of LDKT
* Prior participation in a transplant HC
* Prior or current participation in the NKF PM program

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2022-12-18 (Actual)

PRIMARY OUTCOMES:
Live donor kidney transplants | 1 Year Post-Intervention
  The primary outcome for this study is the proportion of enrolled patients with live donor kidney transplants after 1 year.

SECONDARY OUTCOMES:
Live donor evaluations | 1 Year Post-Intervention
  A secondary outcome for the study is the proportion of enrolled patients with a live donor evaluation at the one-year endpoint. A live donor evaluation is defined as the completion of a transplant evaluation to determine whether a potential living donor is eligible to donate.
Live donor inquiries | 1 Year Post-Intervention
  A secondary outcome for the study is proportion of enrolled patients with live donor inquiries at the one-year endpoint. A live donor inquiry is when an individual contacts the transplant center to express interest in living donation, regardless of when they complete the entire live donor evaluation.

OTHER OUTCOMES:
Improvement in live donor kidney transplant knowledge measured through Living Donation Kidney Transplant Knowledge (LDKT-K) scale score | Baseline, 1 Week Post-Intervention, 6 Weeks Post-Intervention, and 12 Weeks Post-Intervention
  An improvement in patient knowledge is measured by the change in score of a scored instrument, the Living Donation Kidney Transplant Knowledge Scale (LDKT-K). The LDKT-K is a scored true or false questionnaire that tests patient's knowledge on living donation. A higher score indicates that a participant answered more questions correctly.
Improvement in live donor kidney transplant readiness measured through Living Donation Kidney Transplant Readiness scale (LDKT-R) score | Baseline, 1 Week Post-Intervention, 6 Weeks Post-Intervention, and 12 Weeks Post-Intervention
  Improvement in patient readiness to pursue LDKT is measured by a scored instrument, the Living Donation Kidney Transplant Readiness Scale (LDKT-R). The LDKT-R is a 5-point scale where patient's self report their readiness to pursue living donation and where in the process they are (i.e., they are beginning to think about living donation, have spoken with potential donors, etc.) A higher score on this assessment indicates greater readiness to pursue LDKT.
Reduced health care mistrust measured through Health Care Distrust Scale (HCDS) score | Baseline, 1 Week Post-Intervention, 6 Weeks Post-Intervention, and 12 Weeks Post-Intervention
  Reduction in patient mistrust towards the health care system is measured through a scale, the Health Care Distrust Scale (HCDS). This scale is a 5-point Likert scale that measures the degree of agreement patients have on statements regarding their trust of the medical system. For example, one such statement reads "the health care systems lie to make money." A higher score on this assessment indicates higher levels of mistrust of the health care system.
Reduced live donor kidney transplant concerns measured through measured Living Donation Kidney Transplant Concerns scale (LDKT-C) score | Baseline, 1 Week Post-Intervention, 6 Weeks Post-Intervention, and 12 Weeks Post-Intervention
  Patient's concerns towards LDKT is measured using a 5-point scale, the Living Donation Kidney Transplant Concerns scale (LDKT-C) where patients indicate their level of concern towards common concerns patients have regarding living donation. A higher score on this assessment indicates higher levels of concern towards living donation.
Greater amount of time spent discussing LDKT and higher quality interactions measured through the Talking About Living Donation (TaLKeD) instrument | Baseline, 1 Week Post-Intervention, 6 Weeks Post-Intervention, and 12 Weeks Post-Intervention
  The time patients speak with others about LDKT and whether these interactions are of higher quality compared to pre-intervention is measured through a self-report instrument, Talking About Living Donation (TaLKeD), that asks the cumulative time patient's spoke with others (family, friends, etc.) about living donation and their perceived quality of these interactions (poor, fair, good, very good, excellent).
Improvement in self-efficacy discussing LDKT measured through Living Donation Kidney Transplant Self-Efficacy scale (LDKT-SE) score | Baseline, 1 Week Post-Intervention, 6 Weeks Post-Intervention, and 12 Weeks Post-Intervention
  Patient's self-efficacy towards doing activities to pursue LDKT (e.g. willingness and confidence to approach others for donation, following-up with potential donors) is measured through a self-report instrument, the Living Donation Kidney Transplant Self-Efficacy (LDKT-SE) scale. A higher score on this assessment indicates higher self-efficacy for patients pursuing LDKT.

CONTACTS AND LOCATIONS:
Overall Officials: James R Rodrigue, Ph.D., Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Undecided